CLINICAL TRIAL: NCT05794659
Title: A Randomized Phase 2 Study to Evaluate the Efficacy and Safety for Adjuvant Therapeutic Cancer Vaccine (AST-201, pUMVC3-hIGFBP-2) in Patients With Advanced Ovarian Cancer (Cornerstone-004)
Brief Title: Adjuvant Therapeutic Cancer Vaccine (AST-201, pUMVC3-hIGFBP-2) in Patients With Advanced Ovarian Cancer
Acronym: Cornerstone4
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aston Sci. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PN-201-22
Record Dates: First submitted 2023-03-07; First posted 2023-04-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Advanced Ovarian Cancer
Keywords: cancer vaccine; phase 2 study; Advanced ovarian cancer; homologous-recombination proficient (HRP)
MeSH Terms: interventions — Paclitaxel; Carboplatin; Saline Solution; sargramostim

STUDY DESIGN:
Intervention Model Description: Single blind, randomized, placebo-controlled, multicenter, phase 2 clinical study
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AST-301 (Experimental): AST-201 with rhuGM-CSF (3-week interval, 3 cycles in total)
  Standard chemotherapy (paclitaxel/carboplatin) (3-week interval, 6 cycles in total)
  * Both AST-201/rhuGM-CSF or Placebo/rhuGM-CSF will be given intradermally 2 weeks after each combination chemotherapy (on Day 15 of each cycle) for 3 cycles
  Interventions: Biological: AST-201; Drug: Paclitaxel; Drug: Carboplatin; Drug: rhuGM-CSF(Granulocyte-Macrophage Colony-Stimulating Factor)
- Placebo (Placebo Comparator): Placebo with rhuGM-CSF (3-week interval, 3 cycles in total)
  Standard chemotherapy (paclitaxel/carboplatin) (3-week interval, 6 cycles in total)
  *Both AST-201/rhuGM-CSF or Placebo/rhuGM-CSF will be given intradermally 2 weeks after each combination chemotherapy (on Day 15 of each cycle) for 3 cycles
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Placebo; Drug: rhuGM-CSF(Granulocyte-Macrophage Colony-Stimulating Factor)

INTERVENTIONS:
Biological: AST-201 — i.d. (3-week interval, 3 cycles in total)
  Other Names: pUMVC3-hIGFBP-2 multi-epitope plasmid DNA vaccine
  Arms: AST-301
Drug: Paclitaxel — 3-week interval, 6 cycles in total
  Other Names: Taxol
Drug: Carboplatin — 3-week interval, 6 cycles in total
  Other Names: Paraplatin
Drug: Placebo — i.d. (3-week interval, 3 cycles in total)
  Other Names: Normal saline (USP)
  Arms: Placebo
Drug: rhuGM-CSF(Granulocyte-Macrophage Colony-Stimulating Factor) — i.d. (3-week interval, 3 cycles in total)
  Other Names: sargramostim; Leukine

SUMMARY:
The purpose of this phase 2 study is to assess the efficacy and safety for adjuvant therapeutic cancer vaccine AST-201 (pUMVC3-hIGFBP-2) in patients with newly diagnosed homologous-recombination proficient(HRP) advanced ovarian cancer (Stage III) after debulking surgery. Patients will receive AST-201 with rhuGM-CSF(Colony Stimulating Factor) or placebo with rhuGM-CSF in combination with standard adjuvant chemotherapy(Paclitaxel/Carboplatin).

DETAILED DESCRIPTION:
The study will comprise a screening period of -28 Days prior to initiation of study treatment (Day 1); an enrollment period of 24 months; the treatment duration will be approximately of 5 months.

The study will evaluate whether the addition of AST-201/rhuGM-CSF to the standard adjuvant chemotherapy will extend the Progression Free Survival(PFS) rate. Survival follow-up will be performed every 3 months (±14 days) after the End of treatment (EOT) visit for 2 years after randomization and every 6 months (±28 days) thereafter until disease progression or death from any cause or withdrawal of consent whichever comes first. Survival follow-up visits will be conducted by telephone, in-person visit, or chart review. The end of study (EOS) is defined as 2 years after the date of last patient enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage III (FIGO classification) epithelial ovarian cancer including primary peritoneal cancer, fallopian-tube cancer
* Has received upfront surgery and optimally debulked(a residual tumor less than 1 cm)
* Can start adjuvant therapy within 6 weeks of debulking surgery
* Has Homologous Recombination Proficiency (HRP) tumor defined by FDA-approved testing
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Demonstrates adequate organ function.

Exclusion Criteria:

* Has a history of hypersensitivity or other contraindications to rhuGM-CSF
* Has a history of active malignancy ≤5 years prior to first administration of investigational drug except for adequately treated non-melanoma skin cancer or epithelial carcinoma without evidence of disease
* Is on immune suppression therapy or has a history of immune suppression therapy ≤4 weeks prior to the first administration of investigational drugs
* Has active or prior autoimmune disease or inflammatory disease
* Has active infectious disease including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | overall study duration (approximately 48 months)
  the time from the date of randomization to disease progression, or death from any cause whichever occurs first

SECONDARY OUTCOMES:
2-year PFS rate | 24months from the first dose of AST-301 administration
  proportion of patients alive without disease progression or death at two years after the randomization
Overall Survival (OS) | overall study duration (approximately 48 months)
  the time from the date of randomization to death from any cause
AST-201 specific immunogenicity by Interferon gamma (IFN-gamma) enzyme-linked immunospot (ELISpot ) | 17months
  AST-201 specific IFN-gamma ELISpot
Number of participants with Adverse events as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0) | 5 months
  Adverse events (AEs) Treatment-emergent adverse events (TEAEs) Serious adverse events (SAEs) Vital signs Physical examination Eastern Cooperative Oncology Group (ECOG) performance status Electrocardiogram (ECG) test Laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Hyunwon Shin, MD, PhD, Study Director — hyunwon.shin@astonsci.com
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No